CLINICAL TRIAL: NCT02895022
Title: Determination of ED95 of 2% Lidocaine With Epinephrine for Converting Analgesia Epidural Anesthesia in Surgical Epidural in the Labor Current Cesarean
Brief Title: EpiConCES - Epidural Lidocaine for Conversion to CaEsarean Section
Acronym: EpiConCES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0271; 2016-000224-26 (Other: 2016-000224-26)
Record Dates: First submitted 2016-07-04; First posted 2016-09-09 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Pregnant Women>37SA
MeSH Terms: interventions — Lidocaine; Cesarean Section

ARMS (1):
- Lidocaine 2% adrénalinée (Experimental): The main objective is to determine the ED95 dose of 2% lidocaine with epinephrine injected into the epidural catheter for which it does not arise from failure to surgical anesthesia for cesarean during labor.
  Interventions: Drug: Lidocaine 2% adrénalinée; Device: Epidural catheter; Procedure: Caesarean section

INTERVENTIONS:
Drug: Lidocaine 2% adrénalinée
Device: Epidural catheter
Procedure: Caesarean section

SUMMARY:
The need to resort to a midwifery course work in cesarean is a common practice. Epidural analgesia for labor analgesia is practiced in 90% of women in obstetric work, as when the cesarean decision is taken course work in practice and the recommendations are to use the epidural catheter in place to convert the epidural analgesia in epidural anesthesia by re-injecting a local anesthetic on the catheter. General anesthesia is reserved only cases of extreme urgency and cons-indications for regional anesthesia as a purveyor of high maternal morbidity and mortality.

The initial assumption is that the 2% lidocaine with epinephrine is the optimal and recommended local anesthetic solution.

DETAILED DESCRIPTION:
There is a real variability in the volume administered by practitioners repository fault.

The main objective is to determine the ED95 dose of 2% lidocaine with epinephrine injected into the epidural catheter for which it does not arise from failure to surgical anesthesia for cesarean during labor.

The secondary objectives are to determine the failure risk factors, the hemodynamic consequences related to the volume administered and evaluate maternal satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant > 37SA
* Between 150 and 190cm
* IMC between 20 and 40
* Single pregnancy
* Elective cesarean indication during obstetric labor

Exclusion Criteria:

* Presentation of siege
* Extreme and semi emergency caesarean indication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-09-05 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Success or failure of lidocaine 2% with epinephrine dose administered | at day 1

SECONDARY OUTCOMES:
Study tolerance of epidural anesthesia for caesarean section | at day 1
  Study tolerance - including hemodynamics - of epidural anesthesia for caesarean section depending on the dose of 2% lidocaine with epinephrine administered.
maternal pain (Visual Analog Scale) | at day 1
maternal satisfaction | at day 1
nausea and vomiting intraoperatively | at day 1
blood pressure (PAM, PAS (mmHg)) | at day 1
fluid replacement (ml) | at day 1
hypotension | at day 1
necessary to use vasopressors | at day 1
Apgar score | at day 1
fetal arterial and venous cord pH | at day 1
Intravenous sedation for inadequate anesthesia | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Martine BONNIN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France